CLINICAL TRIAL: NCT00352911
Title: A Randomized, Placebo-controlled, Dose Escalating, Phase II Trial of the Anti -HIV-Activity and Safety of VGX-410 (Mifepristone) in HIV-1 Infected Subjects
Brief Title: Antiviral Activity and Safety of Mifepristone at 2 Doses in HIV-1 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VGX Pharmaceuticals, LLC (Industry)
Responsible Party: VGX Pharmaceuticals, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VT004
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: HIV Infections
Keywords: HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Mifepristone

ARMS (2):
- VGX-410 (Mifepristone) (Active Comparator): 150mg twice daily of VGX-410 for 14 days and, if well tolerated, a dose escalation to 300mg twice daily of VGX-410 for 14 days
  Interventions: Drug: VGX-410 (Mifepristone)
- Placebo for VGX-410 (Mifepristone) (Placebo Comparator): 150mg twice daily of placebo for VGX-410 for 14 days and, if well tolerated, a dose escalation to 300mg twice daily of placebo for VGX-410 for 14 days
  Interventions: Drug: Placebo for VGX-410 (Mifepristone)

INTERVENTIONS:
Drug: VGX-410 (Mifepristone)
  Other Names: Mifeprex
  Arms: VGX-410 (Mifepristone)
Drug: Placebo for VGX-410 (Mifepristone)
  Arms: Placebo for VGX-410 (Mifepristone)

SUMMARY:
The objective of the study is to determine whether mifepristone (VGX-410) has anti-HIV-1 activity at doses of either 300 mg or 600 mg per day after oral administration for 14 days at each dose level.

DETAILED DESCRIPTION:
VT004 is a double-blind, randomized, placebo-controlled Phase II study of two doses of orally administered mifepristone (VGX-410) (300 and 600 mg) taken as a twice daily (BID) dosage (150mg BID and 300mg BID) in a dose-escalating fashion for 14 days at each dose level to determine antiviral activity and safety in HIV-1-infected participants. At entry, 18 subjects will be randomized in a 5:1 fashion (15 on active drug: 3 on placebo) to receive escalating doses of VGX-410 or matching placebo. Patients will be randomized to receive 300 mg (as 150 mg BID dose) of VGX-410 or matching placebo for 14 days. In patients that complete this dose without significant safety concerns or side effects, the dose will be increased to 600 mg (as 300 mg BID dose) or matching placebo for 14 days. Patients must meet all inclusion/exclusion criteria listed below and be seen on a weekly basis by study personnel while on study drug. Patients must return ~ one month after finishing the study therapy for examination and safety labs.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4 cell count > 200
* Plasma HIV-1 RNA > 2000 copies/mL and have not received antiretroviral therapy within the 16 weeks prior to entry
* Absolute neutrophil count > 750/mm3
* Hemoglobin > 10 g/dL
* Platelet count > 100,000 mm3
* Creatinine < 2 X upper limit of normal [ULN] (fasting)
* AST (SGOT), ALT (SGPT), and alkaline phosphatase < 2 X ULN
* Total bilirubin < 2.5 X ULN
* Albumin > 3 g/dL
* Serum lipase < 1.5 X ULN
* Thyroid stimulating hormone (TSH) within normal limits
* Plasma cortisol > 20 mcg/dL, 30 minutes after cosyntropin administration
* Negative pregnancy test and willing to use effective birth control during the study
* Karnofsky performance score > 80 within 30 days prior to study entry
* Men and women >= 18 years of age

Exclusion Criteria:

* Receipt of antiretroviral treatment within the 16 weeks prior to study entry
* Chronic adrenal failure, adrenal insufficiency, personal or family history of autoimmune endocrine disease, history of active hepatitis B or C, or current treatment for hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Presence of diabetes mellitus
* Pregnancy within 90 days prior to study entry or breast-feeding
* Dysfunctional uterine bleeding within the 12 months prior to study entry
* Any current hormonal contraception or intrauterine device (IUD) use
* Use of drugs that are inhibitors or inducers of metabolism by the cytochrome P450 3A4 within 7 days prior to study entry
* Use of systemic corticosteroids or hormonal agents within 90 days prior to study entry
* Use of any immunomodulator, HIV vaccines, or investigational therapy within 90 days prior to study entry
* Any vaccination within 30 days prior to study entry
* Use of systemic cytotoxic chemotherapy within 90 days prior to study entry
* History of allergy to mifepristone or its formulations
* Active drug or alcohol use
* Serious illness requiring systemic treatment and/or hospitalization for at least 14 days prior to study entry
* Weight < 40 kg or 88 lbs. within 90 days prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Princy Kumar, M.D., Principal Investigator — Georgetown University; Valerianna Amorosa, MD, Principal Investigator — Veteran's Hospital of Philadelphia; Pablo Tebas, M.D., Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Veterans Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- VGX-410 (Mifepristone); Placebo for VGX-410 (Mifepristone): 150mg twice daily for 14 days and if well tolerated, dose escalation to 300mg twice daily for 14 days
Period: 150mg Twice Daily (14 Days)
Arm/Group | VGX-410 (Mifepristone) | Placebo for VGX-410 (Mifepristone)
Started | 16 | 3
Completed | 16 | 3
Not Completed | 0 | 0
Period: 300mg Twice Daily (14 Days)
Arm/Group | VGX-410 (Mifepristone) | Placebo for VGX-410 (Mifepristone)
Started | 16 | 3
Completed | 15 | 3
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VGX-410 (Mifepristone) | Placebo for VGX-410 (Mifepristone) | Total
Number analyzed (Participants) | 16 | 3 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (8.0) | 37.7 (7.4) | 41.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 14 | 3 | 17
Region of Enrollment [Number; unit: participants]
  United States | 16 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Log Change in Viral Load From Baseline (Day 1) to Day 56
Description: Mean log change in HIV RNA viral load (significant reduction is considered >0.5 log 10) from baseline (Day 1) to Day 56 following 150mg twice daily for 14 days, dose escalation to 300mg twice daily for 14 days and then 28 days off treatment.
Time Frame: Baseline (Day 1) to Day 56
Measure: Log Mean (Standard Deviation); unit: copies/mL on log scale
Arm/Group | VGX-410 (Mifepristone) | Placebo for VGX-410 (Mifepristone)
Number analyzed (Participants) | 16 | 3
copies/mL on log scale | 0.18 (0.28) | 0.42 (0.39)

ADVERSE EVENTS:
Time Frame: AEs that occurred during the treatment period (Days 1-28) of the study.
Arm/Group | VGX-410 (Mifepristone) | Placebo for VGX-410 (Mifepristone)
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/3
Other Adverse Events (participants affected / at risk) | 10/16 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-410 (Mifepristone) (N=16) | Placebo for VGX-410 (Mifepristone) (N=3)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-410 (Mifepristone) (N=16) | Placebo for VGX-410 (Mifepristone) (N=3)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Food Allergy (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Libido Increased (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 | 1
Hot Flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less